CLINICAL TRIAL: NCT04425577
Title: Ultrasound Evaluation Versus Direct Measurement of Uterine Cavity Length: a Prospective Study
Brief Title: Ultrasound Evaluation Versus Direct Measurement of Uterine Cavity Length
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Ashli Lawson, Physician, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001082
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Dysmenorrhea; Heavy Menstrual Bleeding; Contraception
MeSH Terms: conditions — Dysmenorrhea; Menorrhagia

STUDY DESIGN:
Intervention Model Description: Patients who are clinically undergoing intrauterine device (IUD) placement will be consecutively studied
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transabdominal Ultrasound (Other): All patients enrolled will undergo a transabdominal ultrasound at a specified time point as outlined in the protocol.
  Interventions: Diagnostic Test: Transabdominal Ultrasound

INTERVENTIONS:
Diagnostic Test: Transabdominal Ultrasound — Transabdominal Ultrasound

SUMMARY:
To determine if uterine cavity length on transabdominal pelvic ultrasound corresponds to uterine cavity length at time of IUD insertion. If transabdominal pelvic ultrasound is validated as a tool for measuring uterine cavity length, it can be used to guide physicians and subsequently patients in IUD insertion planning.

DETAILED DESCRIPTION:
Levonogesterel (progestin only) IUDs have been used in the adult population for decades and due to their safety and efficacy are now successfully used in the nulliparous and adolescent population for menstrual regulation, dysmenorrhea, and contraception. IUDs have the highest continuation rate among teens of all forms of contraception at 12 months (86%). IUDs reduce menstrual flow by 90% 12 months post insertion, decrease menstrual cramp severity, and have greater than 99% effective contraception. All of this make IUDs an attractive option for our teens and their caregivers

At time of IUD insertion, a uterine sound is used to measure the cavity length. A sound is a rigid instrument that is placed inside the uterus to directly measure the uterine cavity length and is the standard first step prior to IUD insertion. The cavity length will ultimately determine the type and size of IUD that can be placed. Two manufacturers, Mirena ® and Sklya ® are currently being used in clinical practice. Mirena requires uterine cavity length between 6-10 cm and Sklya requires 4-8 cm length. To determine this length requires a pelvic exam and the use of uterine sound, however, approximately 50% of our patient population is unable to tolerate pelvic exams due to a variety of factors, such as developmental disabilities or pain. Thus, this requires patients to go under general anesthesia to have their IUD placed. The goal of this study is to determine if the actual uterine cavity length corresponds to the transabdominal measurement of the uterine cavity length.

Uterine size is largely under the influence of estrogen and as an adolescent progresses through puberty the dimensions of the uterus change. Given that a large portion of families seeking menstrual suppression & regulation present relatively close to menarche (mean age of 12.3 years old) there is a precedent for an institutional standard for pre-IUD insertion transabdominal ultrasound to ensure the uterus is of sufficient caliber

Prior research has focused on those undergoing intra-operative placement of a Mirena IUD. In one retrospective chart review of 56 adolescent patients with developmental disabilities, there was a 3.7% (2/56) failure rate of intra-operative IUD placement (abandoned IUD insertion in the operating room after anesthesia administration). One failure was due to the pelvimetry of the child and the other was due to a uterine cavity length of 4cm which was deemed insufficient for the Mirena IUD. In addition, two other patients had a uterus sound to less than 6 (5cm and 5.5cm) and Mirena was inserted anyways (Skyla was not available). About half of these patients had a pre-operative transabdominal US of the pelvis and the total uterine length was measured with an average length of 8.3cm. All uterine cavities were measured intra-op with an average length of 7.4cm.

Ultimately, all prior research has measured the length of the full uterus (uterine fundus, body of the uterus, and cervix) which is not representative of the measurement in question for IUD placement, the uterine cavity length. We propose a prospective cohort pilot study to compare transabdominal ultrasound measurements with uterine sound measurements to determine uterine cavity length. If these measures correlate, transabdominal US could be a validated pre-insertion tool for the physician and patient to avoid unnecessary anesthetic events and have appropriate IUDs available for insertion.

ELIGIBILITY:
Inclusion Criteria:

* Females age 12 - 22 years old at time of transabdominal ultrasound whom are being considered for IUD placement as part of routine clinical care will be approached for inclusion in the study.
* IUD inserted between 12/1/19 and 12/1/20
* Received a transabdominal US of the uterus

Exclusion Criteria:

* US never performed
* Mullerian anomaly

Ages: 12 Years to 22 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — This is for intrauterine device placement so all participants must have a uterus.
Enrollment: 42 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Quantify Temporal Relationship between Transabdominal Ultrasound and Uterine Sound | Within 60 days of enrollment
  To determine if uterine cavity length on ultrasound corresponds to uterine cavity length at time of IUD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Ashli Lawson, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Julie Strickland, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Usinger KM, Gola SB, Weis M, Smaldone A. Intrauterine Contraception Continuation in Adolescents and Young Women: A Systematic Review. J Pediatr Adolesc Gynecol. 2016 Dec;29(6):659-667. doi: 10.1016/j.jpag.2016.06.007. Epub 2016 Jul 4. PMID 27386754
- [Background] Savasi I, Jayasinghe K, Moore P, Jayasinghe Y, Grover SR. Complication rates associated with levonorgestrel intrauterine system use in adolescents with developmental disabilities. J Pediatr Adolesc Gynecol. 2014 Feb;27(1):25-8. doi: 10.1016/j.jpag.2013.08.010. Epub 2013 Dec 4. PMID 24315712
- [Background] Dizon CD, Allen LM, Ornstein MP. Menstrual and contraceptive issues among young women with developmental delay: a retrospective review of cases at the Hospital for Sick Children, Toronto. J Pediatr Adolesc Gynecol. 2005 Jun;18(3):157-62. doi: 10.1016/j.jpag.2005.03.002. PMID 15970247
- [Background] Lacy J. Clinic opinions regarding IUCD use in adolescents. J Pediatr Adolesc Gynecol. 2006 Aug;19(4):301-3. doi: 10.1016/j.jpag.2006.05.013. No abstract available. PMID 16873036